CLINICAL TRIAL: NCT06635551
Title: Comparison of Vascular Catheter-Related Thrombosis and Risk Factors Using Daily Bedside Ultrasonography After Oncologic and Non-Oncologic Major Surgery
Brief Title: Comparison of Vascular Catheter-Related Thrombosis and Risk Factors After Oncologic and Non-Oncologic Major Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Assistant Prof Levent Özdemir, M.D., Assistant Professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/555
Record Dates: First submitted 2024-08-21; First posted 2024-10-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-12

CONDITIONS: Catheter Related Complication; Thromboses, Venous; Surgery
Keywords: Central Venous Catheters; Venous Thrombosis; Ultrasonography
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Catheter-related thrombosis in oncologic patients after major surgery (Experimental): Cancer patients who will receive central venous catheter
  Interventions: Diagnostic Test: Ultrasonographic evaluation of vascular catheter-related thrombosis after oncological surgery.
- Catheter-related thrombosis in non-oncologic patients after major surgery (Active Comparator): Patients without known cancer who will receive a central venous catheter
  Interventions: Diagnostic Test: Ultrasonographic evaluation of vascular catheter-related thrombosis after non-oncological surgery.

INTERVENTIONS:
Diagnostic Test: Ultrasonographic evaluation of vascular catheter-related thrombosis after oncological surgery. — In patients who will undergo oncological surgery and have a central venous catheter, the presence of thrombosis, its duration of occurrence and its dimensions will be evaluated by ultrasonography.
  Arms: Catheter-related thrombosis in oncologic patients after major surgery
Diagnostic Test: Ultrasonographic evaluation of vascular catheter-related thrombosis after non-oncological surgery. — In patients who will undergo non-oncological surgery and have a central venous catheter, the presence of thrombosis, its duration of occurrence and its dimensions will be evaluated by ultrasonography.
  Arms: Catheter-related thrombosis in non-oncologic patients after major surgery

SUMMARY:
The aim of this study was to prospectively evaluate vascular catheter-related thrombosis and risk factors using daily bedside ultrasonography after oncologic and non-oncologic major surgery.

DETAILED DESCRIPTION:
Vascular catheters (VC) are one of the most frequently performed interventional procedures in both critically ill patients in intensive care units and patients scheduled for major surgery. Recognition of VC-related complications has increased in recent years, and among them, VC-related thrombosis (VCRT) is frequently seen. The reported incidence of VCRT is variable, up to an overall rate of 14-40% for symptomatic events, and may result in pulmonary embolism. Ultrasonography is used frequently and effectively to diagnose intravascular thrombosis and occlusion and provide early intervention. It has been observed that the diagnosis of VCRT can usually be made just before VC is removed or when it becomes symptomatic. Because venous thrombosis formation is a result of altered blood flow, vascular endothelial damage, or altered blood structure, VCRT can occur very early because certain risk factors are present at the time of catheterization. The evolution of VCRT may differ from classic deep vein thrombosis (DVT) depending on existing or removed catheter- or patient-related risk factors. Although there are studies in intensive care patients, the clinical significance of VCRT in patients scheduled for major surgery has not yet been clarified. The time from the first day of catheter placement to the onset of VCRT is not clearly known, and the evolution of VCRT size over time before and after VC removal has not been evaluated. For this reason, it was aimed to evaluate VCRT with ultrasound on a daily basis in the period from insertion to removal of the VC and to evaluate it with a prospective study design in order to detect possible risk factors. Adult patients who will undergo major surgery under elective conditions and are planned to have a central venous catheter inserted will be included in the study. Patients who are decided to have VC implanted will be checked for any thrombus in the vascular structure using ultrasound (US) before the procedure is performed. VC size and length, insertion site, and use of ultrasound guidance will be recorded. Ultrasound detection of VCRT is planned to be performed daily before VC insertion and until VC is removed or the patient is discharged from the intensive care unit. If there is no thrombus between the insertion of the VC and the removal of the VC or until the patient is discharged, patients will be considered as having not developed VCRT. When VCRT is detected, the decision to leave or remove the catheter or initiate therapeutic anticoagulation will be made independently by the patient's responsible physician. A linear probe will be used for ultrasound diagnostic imaging of catheter-related thrombosis. Patients will be examined in the supine position. Doppler ultrasound will be used to evaluate the internal jugular (IJV), subclavian (SCV), femoral (FV), or axillary vein on the same side as the IJV. Ultrasound criteria for the diagnosis of VCRT will require the presence of at least two of the following: intravenous echogenic filling defect, lack of compression of the vein, or abnormal color Doppler pattern. The thrombosis size will be evaluated as follows: In the axial plane, the section with the largest thrombosis area will be selected to measure the maximum and minimum distances, and the maximum distance will be defined as the diameter of the thrombosis. In the longitudinal plane, the length of the thrombosis will be measured. The ultrasound will be performed by an experienced specialist who is competent in bedside ultrasound and is not responsible for patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18-80 years old)
* No hematological disease causing hypercoagulability
* Not receiving anticoagulant/antifibrinolytic medications at the therapy dose
* The vascular structure can be visualized with US
* No thrombosis in the US control before catheter placement
* The catheter is not inserted for renal replacement therapy

Exclusion Criteria:

* Presence of renal failure
* Pediatric patients
* Presence of hematological malignancy
* Inadequate US imaging

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of catheter related vascular thrombosis after surgery | The vascular catheter will be monitored for the duration of its stay, at least 10 days if possible.
  The incidence of vascular catheter-related thrombus in oncologic and non-oncologic surgery patients.

SECONDARY OUTCOMES:
Time from vascular catheter placement to the onset of thrombus formation | Daily assessment until vascular catheter removal, if possible for at least 10 days postoperatively
  The time from the placement of the vascular catheter until the first detection of thrombus according to US criteria
Relationship between demographic characteristics of patients (age, gender and additional diseases) recorded on the preoperative anesthesia assessment form and vascular catheter-related thrombosis | From preoperative anesthesia assessment to postoperative day 10
  Comparison of patients according to gender, age and additional diseases
Daily changes in thrombus area (cm2) from the diagnosis of vascular catheter-related thrombus to catheter removal or patient discharge | Daily assessment until vascular catheter removal, if possible for at least 10 days postoperatively
  Daily US evaluation of the area in patients with catheter related thrombus formation
The incidence of severe complications such as pulmonary embolism, cerebrovascular disease or acute coronary ischemia that may occur due to vascular catheter-related thrombosis | Daily assessment until vascular catheter removal, if possible for at least 30 days postoperatively
  Evaluation for the development of pulmonary embolism, cerebrovascular occlusions and acute coronary ischemia
Lenght of stay at hospital/ICU and mortality | From date of surgery until the date of discharge of patient or date of death from any cause, whichever came first, assessed up to 10 weeks
  To compare the length of hospital stay of patients with and without catheter-related thrombus and to determine mortality rates.

CONTACTS AND LOCATIONS:
Overall Officials: Levent Özdemir, Principal Investigator — Mersin University, Faculty of Medicine, Mersin, Turkiye
Locations (1):
- Mersin University, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Timsit JF, Rupp M, Bouza E, Chopra V, Karpanen T, Laupland K, Lisboa T, Mermel L, Mimoz O, Parienti JJ, Poulakou G, Souweine B, Zingg W. A state of the art review on optimal practices to prevent, recognize, and manage complications associated with intravascular devices in the critically ill. Intensive Care Med. 2018 Jun;44(6):742-759. doi: 10.1007/s00134-018-5212-y. Epub 2018 May 12. PMID 29754308
- [Background] Wu C, Zhang M, Gu W, Wang C, Zheng X, Zhang J, Zhang X, Lv S, He X, Shen X, Wei W, Wang G, Lu Y, Chen Q, Shan R, Wang L, Wu F, Shen T, Shao X, Cai J, Tao F, Cai H, Lu Q; Study Group of Central Venous Catheter-related Thrombosis. Daily point-of-care ultrasound-assessment of central venous catheter-related thrombosis in critically ill patients: a prospective multicenter study. Intensive Care Med. 2023 Apr;49(4):401-410. doi: 10.1007/s00134-023-07006-x. Epub 2023 Mar 9. PMID 36892598
- [Background] Debourdeau P, Lamblin A, Debourdeau T, Marcy PY, Vazquez L. Venous thromboembolism associated with central venous catheters in patients with cancer: From pathophysiology to thromboprophylaxis, areas for future studies. J Thromb Haemost. 2021 Nov;19(11):2659-2673. doi: 10.1111/jth.15487. Epub 2021 Aug 26. PMID 34363736